CLINICAL TRIAL: NCT05593406
Title: The Effect of Mechanical Vibration on Spasticity and Balance in Children With Cerebral Palsy
Brief Title: Mechanical Vibration on Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: Thomas Besios (Unknown); Georgios Paras (Unknown); Konstantinos Chandolias (Unknown)
Responsible Party: Principal Investigator, Aourela Gkioni, Msc Cand Aourela Gkioni, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: AG12071996
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Cerebral Palsy; Spastic Hemiplegic Cerebral Palsy
Keywords: Cerebral palsy; Balance; Neurodevelopmental treatment; Whole body vibration; Spasticity
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The children who participated in the study were randomly divided through folders into an intervention group and a control group. The control group continued the physical therapy program they were already following, while the intervention group, in addition to the conventional physical therapy they received, did also receive mechanical vibration.
Who Masked: Participant
Masking Description: Randomly divided through folders
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibration Group (Experimental): The intervention-vibration group, in addition to the conventional physical therapy- NDT they received, were also included in mechanical vibration.
  Interventions: Device: Vibration Group
- Control Group (Active Comparator): The Control group received only conventional physical therapy- NDT.
  Interventions: Other: Control Group

INTERVENTIONS:
Device: Vibration Group — Whole body vibration for 15 minutes in squat and lunge position.
  Other Names: Mechanical Vibration; Neurodevelopmental treatment
  Arms: Vibration Group
Other: Control Group — NDT treatment 2 sessions per week
  Other Names: Neurodevelopmental Treatment
  Arms: Control Group

SUMMARY:
The purpose of this study was to assess the effect of mechanical vibration on spasticity and balance in children with cerebral palsy. The participants of the clinical study are 13 children with CP and age 4-17 years, with a diagnosis of spastic hemiplegic cerebral palsy. More specifically, the participants were randomly divided into a control group and an intervention group, with the first group continuing conventional physical therapy, while the experimental group outside the physical therapy program did also receive mechanical vibration using a hybervibe G10 vibration platform (lasting 15 minutes). The intervention lasted 8 weeks and participants were assessed before the start of the intervention (T1), 1 month after the first assessment (T2) and rechecked 1 month (T3) after the completion of the program using valid and reliable tools.

DETAILED DESCRIPTION:
This is a randomized clinical study and 13 children, aged 4-17 with diagnosed spastic hemiplegic cerebral palsy participated in the research. The collection of the sample and the recording of the data took place in Pediatric Physiotherapy Private Practice centers in Lamia, Trikala and Katerini. Sampling was completed after written consent of the children's parents, as long as they were fully informed about the purposes of the research, the private physical therapy centers and the Human Performance & Rehabilitation Laboratory of the University of Thessaly.

The time period that the clinical study intervention lasted was 8 weeks. The children who participated in the study were randomly divided through folders into an intervention group and a control group. The control group continued the physical therapy program they were already following, while the intervention group, in addition to the conventional physical therapy they received, did also resceive mechanical vibration. The program they were already following was based on the Bobath NDT Neuroevolutionary Method, where, through special manipulations, the emphasis is placed on improving the quality of movement and the functionality of the children, as well as the inclusion of the family in the wider treatment is considered important.

The inclusion of mechanical vibration in the children was carried out in parallel with the conventional physical therapy program they followed. The protocol with the appropriate exercises to be followed on the HyperVibe G10 mini vibration platform had a duration of 15 minutes, with a 2 minute break, the frequency of the mechanical vibration was 14Hz, the opening of the legs (amplitude) on the platform and the range of bending the knees depended on each participant and how safe they felt during the procedure. In front of them there was the possibility of supporting the upper limbs, for a possible loss of balance or if they felt insecure.

ELIGIBILITY:
Inclusion Criteria:

* The children from 4 - 17 years old
* diagnosis of spastic hemiplegic cerebral palsy
* ability to understand simple commands.
* up to level GMFCS III,
* able to stand and walk (with or without mobility aids).

Exclusion Criteria:

* children who have been injected with botulinum toxin up to 3 months before
* children who have undergone selective rhizotomy surgery up to 1 year before,
* uncontrolled epilepsy,
* other pathologies that will affect the outcome of the intervention.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
TUG | 2 months
  TIMED UP AND GO (Scale to asses speed) (the minimum time the better)
PBS | 2 months
  PAEDIATRIC BALANCE SCALE (BERG BALANNCE SCALE MODIFIED) (Scale for assess the balance) (score 0-56)
MAS | 2 months
  Modified Asworth scale (spasticity)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Thessaly, Lamia, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Ahlborg, L., Andersson, C., & Julin, P. (2006). Whole-body vibration training compared with resistance training: Effect on spasticity, muscle strength and motor performance in adults with cerebral palsy. Journal of Rehabilitation Medicine, 38(5). https://doi.org/10.1080/16501970600680262 2. Ahmadizadeh, Z., Khalili, M. A., Ghalam, M. S., & Mokhlesin, M. (2019). Effect of whole body vibration with stretching exercise on active and passive range of motion in lower extremities in children with cerebral palsy: A randomized clinical trial. Iranian Journal of Pediatrics, 29(5). https://doi.org/10.5812/ijp.84436 3. Alashram, A. R., Padua, E., & Annino, G. (2019). Effects of Whole-Body Vibration on Motor Impairments in Patients With Neurological Disorders. In American Journal of Physical Medicine and Rehabilitation (Vol. 98, Issue 12). https://doi.org/10.1097/PHM.0000000000001252 4. Ali, M. S., Awad, A. S., & Elassal, M. I. (2019). The effect of two therapeutic interventions on balance in children with spastic cerebral palsy: A comparative study. Journal of Taibah University Medical Sciences, 14(4). https://doi.org/10.1016/j.jtumed.2019.05.005 5. Andrew Harb and Stephen Kishner. (2022). Modified Ashworth Scale. StatPearls. 6. Bax, M., Goldstein, M., Rosenbaum, P., Leviton, A., Paneth, N., & Dan, B. et al. (2005). Proposed definition and classification of cerebral palsy, April 2005. Developmental Medicine & Child Neurology, 47(8), 571-576. doi: 10.1017/s001216220500112x 7. Cans, C., Dolk, H., Platt, M. J., Colver, A., Prasauskiene, A., & Krägel-Oh-Mann, I. (2007). Recommendations from the SCPE collaborative group for defining and classifying cerebral palsy. Developmental Medicine and Child Neurology, 49(SUPPL. 2). https://doi.org/10.1111/j.1469-8749.2007.tb12626.x 8. Cheng, H. Y. K., Ju, Y. Y., Chen, C. L., Chuang, L. L., & Cheng, C. H. (2015). Effects of whole body vibration on spasticity and lower extremity function in children with cerebral palsy. Human Movement Science, 39. https://doi.org/10.1016/j.humov.2014.11.003 9. Christopher, A., Kraft, E., Olenick, H., Kiesling, R., & Doty, A. (2021). The reliability and validity of the Timed Up and Go as a clinical tool in individuals with and without disabilities across a lifespan: a systematic review: Psychometric properties of the Timed Up and Go. In Disability and Rehabilitation (Vol. 43, Issue 13). https://doi.org/10.1080/09638288.2019.1682066 10. El-Shamy, S. M. (2014). Effect of whole-body vibration on muscle strength and balance in diplegic cerebral palsy: A randomized controlled trial. American Journal of Physical Medicine and Rehabilitation, 93(2). https://doi.org/10.1097/PHM.0b013e3182a541a4 11. Franjoine, M., Darr, N., Held, S., Kott, K., & Young, B. (2010). The Performance of Children Developing Typically on the Pediatric Balance Scale. Pediatric Physical Therapy, 22(4), 350-359. https://doi.org/10.1097/pep.0b013e3181f9d5eb 12. Fratini, A., Bonci, T., & Bull, A. M. J. (2016). Whole body vibration treatments in postmenopausal women can improve bone mineral density: Results of a stimulus focussed meta-analysis. PLoS ONE, 11(12). https://doi.org/10.1371/journal.pone.0166774